CLINICAL TRIAL: NCT01905254
Title: Prospective Comparison of Transient Elastography and Mini-laparoscopic Guided Liver Biopsy in Autoimmune Hepatitis
Brief Title: Transient Elastography in Autoimmune Hepatitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Principal Investigator, PD Dr. med. Ulrike Denzer, Attending physician, Universitätsklinikum Hamburg-Eppendorf
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: UKE IRB 2742
Record Dates: First submitted 2013-07-01; First posted 2013-07-23 (Estimated); Results first posted 2015-05-06 (Estimated); Last update posted 2015-05-06 (Estimated); Status verified 2015-05

CONDITIONS: Liver Cirrhosis
Keywords: Transient elastography; mini-laparoscopy; liver biopsy; liver cirrhosis; autoimmune hepatitis
MeSH Terms: conditions — Liver Cirrhosis; Hepatitis, Autoimmune

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Transient elastography and liver biopsy (Other): All patients with Autoimmune hepatitis (AIH) were investigated with Transient Elastography before liver biopsy
  Interventions: Device: Transient elastography (TE); Other: Liver biopsy

INTERVENTIONS:
Device: Transient elastography (TE) — TE and minilaparoscopic guided liver biopsy were performed by physicians blinded to the results the other within a period of less than 3 months.
Other: Liver biopsy — Minilaparoscopic guided liver biopsy was performed within a period of 3 months of Transient Elastography

SUMMARY:
Recent, research has focused on the evaluation of non-invasive methods for the assessment of liver fibrosis in patients with chronic liver disease. Among these methods, transient elastography is the most promising. The method has been investigated mainly in patients with viral hepatitis. Several studies have shown, that the optimal cut-off value of TE for detection of liver cirrhosis by transient elastography is highly dependent on the aetiology of the underlying liver disease. Only a few studies have evaluated the value of transient elastography for patients with autoimmune liver disease and here primarily patients with PBC and PSC. For patients with autoimmune hepatitis the data is limited. We prospectively investigated the diagnostic accuracy of TE in autoimmune hepatitis compared to liver histology with and without inclusion of the macroscopic appearance using mini-laparoscopy

DETAILED DESCRIPTION:
The aim of the current study was to assess the diagnostic performance of transient elastography for the determination of cirrhosis in patients with autoimmune hepatitis compared to the diagnosis of cirrhosis made on Laparoscopic guided liver biopsy. Patients referred for liver biopsy and transient elastography with a clinical diagnosis of AIH followed in the liver clinic of the Department of Gastroenterology at the UKE were prospectively included in the study.

Inclusion criteria were as follows: Confirmed diagnosis of AIH based on the diagnostic criteria revised by the International Autoimmune Hepatitis Group 2008 (20): 1. liver related autoantibodies, 2. hypergammaglobulinaemia, 3.typical histological findings and 4. absence of viral markers. Exclusion criteria were morbid obesity (BMI > 40), ascites, ileus or subileus, peritonitis, pregnancy, extrahepatic cholestasis and a severe inflammatory flare of AIH.

Blood liver tests including gamma-globulines, IgG, IgM, liver related autoantibodies (ANA, AMA, LKM, SMA, SLA) and viral markers (HBsAg, Anti HBs, Anti HBc, Anti HCV, Anti HAV) were performed before LB.

Each patient underwent abdominal ultrasound to exclude extrahepatic cholestasis prior to TE and minilaparoscopic liver biopsy. TE and minilaparoscopy were performed by physicians blinded to the results the other within a period of less than 3 months.

ELIGIBILITY:
Inclusion Criteria:

Confirmed diagnosis of AIH based on the diagnostic criteria revised by the International Autoimmune Hepatitis Group 2008 (20):

1. liver related autoantibodies,
2. hypergammaglobulinaemia,
3. typical histological findings and
4. absence of viral markers.

Exclusion Criteria:

* morbid obesity (BMI > 40),
* ascites, ileus or subileus,
* peritonitis,
* pregnancy,
* extrahepatic cholestasis and
* a severe inflammatory flare of AIH.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2007-08; Primary Completion 2010-08 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ulrike W Denzer, MD, Principal Investigator — Universitätsklinikum Hamburg-Eppendorf; Ansgar W Lohse, MD, Study Chair — Universitätsklinikum Hamburg-Eppendorf
Locations (1):
- Dept of Gastroenterology and Hepatology, University Medical Center Hamburg Eppendorf, Hamburg, Hamburg, Germany

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Thirty-nine patients with AIH were eligible during the study period. Five patients were excluded: 4 patients due to ineffective or incomplete (<60% success rate) liver stiffness measurement, and 1 patient with a severe acute flare of AIH with markedly elevated liver enzymes."
Groups:
- Transient Elastography and Liver Biopsy: Transient elastography was performed by two experienced investigators using a FibroScan (EchoSens, Paris, France), the median value of liver stiffness measurements was recorded in kilopascals (kPa).
  Liver biopsy was carried out within 3 months of TE. Liver biopsies from the right and left lobe were obtained under laparoscopic control using the Tru-cut 16 GAUGE needle (Bard monopty; Bard biopsy systems, Tempe, USA).
  Data analysis was performed on the remaining 34 patients (female: 28 (82%); male: 6 (18 %).
  Indications for liver biopsy and Transient elastography were: 19 patients for follow-up of AIH while receiving immunosuppression and 15 patients for staging and grading of AIH before starting with an immunosuppressive therapy in.
Period: Overall Study
Arm/Group | Transient Elastography and Liver Biopsy
Started | 34
Completed | 34
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Data analysis was performed on 34 patients (female: 28 (82%); male: 6 (18 %). Indications for liver biopsy and Transient elastography were: 19 patients for follow-up of AIH while receiving immunosuppression and 15 patients for staging and grading of AIH before starting with an immunosuppressive therapy in.
Groups:
- Single Arm Study: Alle patients received a liver biopsy and Transient elastopgrapy for follow-up of Autoimmune Hepatitis or staging and grading of Autoimmune hepatitis.
Arm/Group | Single Arm Study
Number analyzed (Participants) | 34
Age, Continuous [Median (Full Range); unit: years] | 53 [21 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 34
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Germany | 34

OUTCOME MEASURES:

1. Primary Outcome: Sensitivity and Specifity of Transient Elastography in Detection of Liver Cirrhosis
Description: The aim of the current study was to assess the diagnostic accuracy (Sens., Spec.) of transient elastography for the determination of cirrhosis in patients with autoimmune hepatitis. TE was compared to the diagnosis of cirrhosis made on histology yielded by laparoscopic guided liver biopsy.
Time Frame: Transient Elastography compared to liver histology
Population: Sensitivity, specifity; Positive and negative predictive value of TE for diagnosis of cirrhosis was analyzed.
Measure: Number; unit: Probability
Groups:
- Transient Elastography in Autoimmune Hepatitis: Liver stiffness (kPa) was correlated to histologic staging of liver cirrhosis
Arm/Group | Transient Elastography in Autoimmune Hepatitis
Number analyzed (Participants) | 34
Probability
  Sensitivity of TE for diagnosis cirrhosis | 0.83
  Specifity of TE for diagnosis cirrhosis | 1.00
  Positive predictive value of TE for cirrhosis | 1.00
  Negative predictive value of TE for cirrhosis | 0.97

ADVERSE EVENTS:
Groups:
- TE in Autoimmune Hepatitis: Alle patients received a liver biopsy and Transient elastopgrapy for follow-up of Autoimmune Hepatitis or staging and grading of Autoimmune hepatitis.
  There were no adverse events.
Arm/Group | TE in Autoimmune Hepatitis
Serious Adverse Events (participants affected / at risk) | 0/34
Other Adverse Events (participants affected / at risk) | 0/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TE in Autoimmune Hepatitis (N=34)
Pain after liver biopsy (Gastrointestinal disorders) | 0
Bleeding after liver biopsy (Hepatobiliary disorders) | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TE in Autoimmune Hepatitis (N=34)
Hypotension (Cardiac disorders) | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes